CLINICAL TRIAL: NCT05240482
Title: Zusanli (ST36) Acupoint Injection With Anisodamine for Postoperative Nausea and Vomiting in Women Following Bariatric Surgery: A Single-center Study
Brief Title: ST36 Acupoint Injection With Anisodamine for Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, hui hou, Principal Investigator, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YX2021-114
Record Dates: First submitted 2022-01-10; First posted 2022-02-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: postoperative nausea and vomiting; bariatric surgery; Zusanli (ST36); anisodamine
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Outcomes will be evaluated by anesthesiologists who are blinded to the treatment allocation. Patients, investigators and observers will be blinded to the patient allocation throughout the entire study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment group (Placebo Comparator): Patients in the placebo group will receive bilateral ST36 injection with normal saline 1ml/point
  Interventions: Procedure: ST36 acupuncture
- ST36 acupoint injection group (Experimental): Patients in the experimental group will receive bilateral ST36 injection with anisodamine 1ml/point
  Interventions: Procedure: ST36 acupuncture

INTERVENTIONS:
Procedure: ST36 acupuncture — ST36 is located on the lateral surface of leg, 3 cun distal to the lower border of the patella, 1 finger-breadth lateral to the anterior crest of the tibia, between the tibialis anterior muscle and the tendon of the extensor digitorum longus. (The breadth of patient's middle finger was the proportional unit of measure "the cun", defined as the distance between the two medial ends of the creases of the interphalangeal joints when the patient's middle finger is flexed).

SUMMARY:
Postoperative nausea and vomiting (PONV) is particularly distressing although it is not a fatal postoperative complication. Numbers of studies have been focused on identifying risk factors and therapies of PONV. Unfortunately, there' no consistent comments for PONV prevention in women after laparoscopic sleeve gastrectomy. Notably, Zusanli (ST36) acupoint and anisodamine have been evidenced to treat various gastrointestinal conditions. The primary outcome of this study was to evaluate the impact of anisodamine injection in ST36 on PONV in women following bariatric surgery.

DETAILED DESCRIPTION:
Acupuncture has been used as a medical technique in China for at least 2,000 years. More recently, it's also been extensively used in managing headache, chronic back pain, and PONV in USA. ST36 acupuncture is reported to be an effective preventive treatment for postoperative nausea and vomiting (PONV). However, It is not clear if it could efficiently prevent PONV in female patient who has underwent bariatric surgery. At the onset of this investigation, we have already identified several methodologic issues, such as the timing of the acupuncture intervention, sample size, perioperative anesthetic techniques, and appropriate control groups. The primary outcome of this study was the total incidence of PONV during the hospital and after the discharge. Participants were randomly assigned into different groups according to the with a computer-generated randomization sequence (http://www.randomization.com). Patients, surgeons, anesthesiologists, nursing staff, and the research assistant, were all blinded to the group assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with an American Society of Anesthesia (ASA) physical status Ⅰ-Ⅲ
2. Scheduled for elective bariatric surgery .

Exclusion Criteria:

1. lack of patient consent
2. patients with contraindications for acupoint injection
3. obesity due to endocrine disorder
4. allergic diathesis for drugs used in the study
5. serious illness (heart, lung, kidney, or liver)
6. coagulation dysfunction
7. pre-existing psychological disorder
8. anticathartic , glucocorticoid or opiates medications

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
The incidence of PONV within the first 24 hours | At 0-24 hours after surgery
  The incidence of PONV within the first 24 hours

SECONDARY OUTCOMES:
Time to the first rescue antiemetics | At 0-24 hours after surgery
  The time from extubation to the first rescue antiemetics
The incidence and severity of PONV assessed at 2, 6, 48, and 72 hours after surgery | At 0-24 hours after surgery
  The incidence and severity of PONV in the anesthesia intensive care unit (AICU) or during the ward.
Early recovery outcomes | Before discharge
  Including the time of first drink, ambulate and flatus
Consumption of propofol | During the surgery
  The consumption of propofol during the surgery
Consumption of remifentanil | During the surgery
  The consumption of remifentanil during the surgery
Consumption of cisatracurium | During the surgery
  The consumption of cisatracurium during the surgery
Consumption of dexmedetomidine | During the surgery
  The consumption of cisatracurium during the surgery
Length of anesthesia | At the end of anesthesia
  From beginning to the end of anesthesia
Length of surgery | At the end of surgery
  From beginning to the end of surgery
Postoperative hospitalization | During hospital
  Days of hospital staying after surgery
QoR-15 | At 24 hours after surgery
  Quality of Recovery-15 (QoR-15) will be used to assess quality of recovery after anesthesia. Total score ranges from 0 to 150. A higher total score means better quality of recovery.
The usage of rescue antiemetic drugs | Within 24 hours after surgery in anesthesia resuscitation unit
  Total usage of rescue antiemetic drugs after surgery
Adverse events | Within 3 months after surgery
  Any adverse events after surgery within postoperative 3 months
BMI | Before surgery and at the postoperative 3 months
  Body mass index
Pittsburgh Sleep Quality Index | Before surgery and at the postoperative 3 months
  Pittsburgh Sleep Quality Index (PSQI) will be assessed the quality of sleep. The higher score means the lower quality of sleep.
Gastrointestinal Symptom Rating Scale | Before surgery and at the postoperative 3 months
  Gastrointestinal symptom rating scale (GSRS) will be used to assess gastrointestinal function. The score ranges from 0 to 45. The higher score means poorer gastrointestinal function .
Hamilton Depression Rating Scale | Before surgery and at the postoperative 3 months
  Hamilton Depression Rating Scale (HAMD) will be used to assess depression. HAMD 24 item version score range 0-96. The higher score means the higher possibility of depression.
Hamilton Anxiety Rating Scale | Before surgery and at the postoperative 3 months
  Hamilton Anxiety Rating Scale (HAM-A) will be used to assess anxiety. Total score ranges from 0 to 56, the higher the score is, the more serious the anxiety is.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Zhang, M.D., Study Chair — The Second Hospital of Anhui Medical University
Locations (1):
- Second Affiliated Hospital of Anhui Medical University, Hefei, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication are to be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will become available when summary data are published.
Access Criteria: Chunxia Huang and Ye Zhang will review requests and criteria to share IPD. Requests are to be sent by email to huangchunxia@ahmu.edu.cn or zhangye_hassan@sina.com.